CLINICAL TRIAL: NCT01751061
Title: Improving Decision Making for Patients With Prolonged Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Pittsburgh (Other); University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00021965; R01HL109823-01A1 (NIH)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Surrogate Decision Makers; Prolonged Mechanical Ventilation
Keywords: prolonged mechanical ventilation; chronic critical illness; decision making; decision aid; decisional support; critical illness; intensive care unit
MeSH Terms: conditions — Critical Illness | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decision aid (Experimental): Web-based decision aid (decision support tool) provided to surrogate decision maker
  Interventions: Behavioral: Decision aid
- Usual care (Active Comparator): usual care in an intensive care unit setting
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Decision aid — A web-based decision aid to assist surrogate decision makers in prolonged mechanical ventilation decisions
  Arms: Decision aid
Other: Usual care — usual ICU care
  Arms: Usual care

SUMMARY:
Deciding about prolonged life support for critically ill patients can be very difficult. Therefore, the investigators are doing a study to see if an internet-based decision aid can improve the quality of decision making for substitute decision makers of patients who are in the intensive care unit (ICU).

DETAILED DESCRIPTION:
The process of making a decision about whether or not to provide prolonged life support is seriously deficient among clinicians and the surrogate decision makers for critically ill patients. To address this problem, we propose a randomized, controlled trial to determine if an innovative web-based decision aid compared to usual care control can improve the quality of decision making (defined as clinician-surrogate concordance for prognosis, quality of communication, and medical comprehension), reduce surrogates' psychological distress (depression, anxiety, and post-traumatic stress syndrome disorder (PTSD) symptoms), and reduce patients' health care costs over 6-month follow up. We will enroll 410 surrogate decision makers for 273 patients (expected average of 1.5 surrogates per patient). This study has the potential both to improve how clinicians and surrogates interact in intensive care units and to increase the likelihood that life support decisions are aligned with patients' values.

ELIGIBILITY:
Inclusion Criteria (Patient characteristics required for surrogate inclusion)

* age ≥18
* ≥10 days of mechanical ventilation interrupted by <96 continuous hours of unassisted breathing (including invasive and non-invasive ventilation)
* no anticipation of imminent (24 hours) death or extubation by the attending.

Exclusion Criteria (Patient characteristics that will exclude surrogates from study enrollment):

* possession of decisional capacity
* no identifiable surrogate, surrogate is unavailable for study procedures such as interviews
* imminent organ transplantation
* chronic neuromuscular disease
* physician refuses permission to approach family and/or patient for consent
* admission for severe burns
* admission for high cervical spine injury
* ventilation for >21 days.

Inclusion criteria for surrogate decision makers:

* age ≥18
* self-identified as participating directly in health care decision making for the incapable patient under relevant state law

Exclusion criteria for surrogate decision makers:

* do not personally know the patient
* need translation assistance because of poor English fluency (the decision aid has not been validated in other languages)
* history of clinically important neurological disorder (e.g., dementia)
* patient dies after meeting inclusion criteria but before surrogates provide consent

Physician and nurse inclusion criteria:

* ICU attending or fellow (physicians) at the time of surrogate enrollment
* bedside ICU nurse present at the time of surrogate enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Cox, MD MPH, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Cox CE, Lewis CL, Hanson LC, Hough CL, Kahn JM, White DB, Song MK, Tulsky JA, Carson SS. Development and pilot testing of a decision aid for surrogates of patients with prolonged mechanical ventilation. Crit Care Med. 2012 Aug;40(8):2327-34. doi: 10.1097/CCM.0b013e3182536a63. PMID 22635048
- [Derived] Cox CE, White DB, Hough CL, Jones DM, Kahn JM, Olsen MK, Lewis CL, Hanson LC, Carson SS. Effects of a Personalized Web-Based Decision Aid for Surrogate Decision Makers of Patients With Prolonged Mechanical Ventilation: A Randomized Clinical Trial. Ann Intern Med. 2019 Mar 5;170(5):285-297. doi: 10.7326/M18-2335. Epub 2019 Jan 29. PMID 30690645

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These numbers reflect primary and secondary surrogate decision makers, not patients, because surrogates were the focus of the trial.
Period: Overall Study
Arm/Group | Decision Aid | Usual Care
Started | 210 | 206
Completed | 154 | 172
Not Completed | 56 | 34
Not completed — Death | 1 | 0
Not completed — patient death | 5 | 0
Not completed — Lost to Follow-up | 40 | 25
Not completed — patient regained decisional capacity | 4 | 8
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Population: primary and secondary surrogate decision makers
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | Usual Care | Total
Number analyzed (Participants) | 210 | 206 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Note that we have broken the population down into primary and secondary surrogate decision makers. However, the two groups sum to the total for intervention and control.
  years
    primary surrogate decision makers: number analyzed (Participants) | 137 | 138 | 275
    primary surrogate decision makers | 49.9 (13.5) | 52.6 (11.6) | 51.2 (12.6)
    secondary surrogate decision makers: number analyzed (Participants) | 73 | 68 | 141
    secondary surrogate decision makers | 46.7 (14.0) | 41.2 (15.4) | 44.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 150 | 297
  Male | 63 | 56 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 198 | 196 | 394
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 2 | 11
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 44 | 25 | 69
  White | 151 | 166 | 317
  More than one race | 2 | 6 | 8
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 210 | 206 | 416

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-surrogate Concordance Scale Score
Description: Concordance is calculated as the absolute value of the difference in prognosis for 1 year patient survival between the surrogate(s) and the clinician (ICU physician), and, therefore, can range from 0 to 100.
  We report pre-intervention to post-intervention difference in the CSCS.
  The CSCS is calculated as the absolute value of the difference between the surrogate's response and that of either the treating ICU physician (primary outcome) or the nurse (secondary outcome) to the question, "What percent chance do you think [the patient/your loved one] has of being alive 1 year from now if the current treatment plan is continued?" Scores can range from 0 to 100 percentage points, and higher values indicate greater discordance.
Time Frame: ~2-7 days post-randomization
Population: Note that the discrepancy between the number of surrogates in these analyses (122 and 127) differs from those enrolled (137 and 138). This is because the CSCS requires complete data at both Interview 1 and Interview 2. Some patients died or regained decisional capacity before Interview 2, leading to loss of surrogates' data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 122 | 127
score on a scale
  Change score | -6.6 [-11.5 to -1.6] | -4.8 [-9.1 to -0.6]
  Interview 1 CSCS score | 33.6 [29.3 to 38.0] | 34.3 [29.9 to 38.8]
  Interview 2 CSCS score | 27.1 [22.8 to 31.4] | 29.5 [25.1 to 33.9]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; We estimated that 210 patients (315 surrogates, assuming ~1.5 per patient) would provide a power of 80% to detect a between-groups mean CSCS score difference of 9 percentage points between Interviews 1 and 2, assuming a baseline mean of 50, SD=24, a type-I error=5%, a correlation between interviews of 0.5, an expectation that 50% of patients would have multiple surrogates, an intraclass correlation coefficient of 0.8 for multiple surrogates for a patient, and 5% dropout before Interview 2; Test type: Superiority — To test the primary hypothesis, we used a general linear model fit with generalized estimating equations, a linear link, and an exchangeable correlation (PROC GENMOD). Model parameters included indictor variables for intervention, Interview 2, the interaction between intervention and Interview 2, and a 4-level site variable. The mean CSCS between-groups difference, corresponding 95% confidence interval (CI), and p value were derived from the intervention-by-Interview 2 interaction term; p < 0.05, GEE — P values were calculated. A two-sided type-I error rate of 0.05 was set for all tests; there were no adjustments for multiple comparisons. All participants were included in analyses as per their group randomization

2. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Total Score
Description: We report here the difference between Interview 1 (baseline) and Interview 4 (6 months post-randomization) for primary surrogate decision makers (not secondary).
  HADS scores can range from 0 to 42 points; higher scores=more distress.
Time Frame: Pre-randomization (study day 1) and 180 days post-randomization
Population: Primary surrogate decision makers only. There is some dropout at 6 months due to patient death.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 101 | 117
units on a scale | -3.8 [-5.3 to -2.3] | -4.0 [-5.1 to -2.8]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; Generalized linear model; Test type: Superiority; p < 0.05, generalized linear model — P values were calculated

3. Secondary Outcome: Post-traumatic Stress Syndrome Inventory
Description: Here we report PTSS score differences between Interview 1 (baseline) and Interview 4 (6 months post-randomization) for primary (not secondary) surrogate decision makers.
  PTSS scores can range from 10-70, with greater scores=more distress.
Time Frame: Pre-randomization (study day 1) and 180 days post-randomization
Population: Primary surrogate decision makers only; there is some dropout at 6 months due to patient death.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 101 | 117
units on a scale | -1.7 [-3.9 to 0.4] | -1.4 [-3.4 to 0.6]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; Test type: Superiority; p < 0.05, generalized linear model — P values were calculated

4. Secondary Outcome: Patient-centeredness of Care Scale
Description: Here we report change in patient-centeredness score between Study day 1 (Interview 1) and 180 days post-randomization (Interview 4) for primary (not secondary) surrogate decision makers.
  Scores can range from 12-48 points, with higher scores=greater patient-centeredness.
Time Frame: Study day 1 and 180 days post-randomization
Population: Primary surrogate decision makers only; there is some dropout at 6 months due to patient death.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 101 | 117
units on a scale | 42.7 [41.3 to 44.1] | 41.8 [40.3 to 43.2]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; Test type: Superiority; p < 0.05, generalized linear models — P values were calculated

5. Secondary Outcome: Medical Comprehension Scale Score
Description: Here we report MCS score differences between Interview 1 (baseline) and Interview 2 (immediately post-intervention) for primary (not secondary) surrogate decision makers.
  Scores can range from 0-8, with greater scores=better comprehension.
Time Frame: Study day 1 (pre-randomization), ~2-7
Population: Note that the discrepancy between the number of surrogates in these analyses (122 and 127) differs from those enrolled (137 and 138). This is because the MCS requires complete data at both Interview 1 and Interview 2. Some patients died or regained decisional capacity before Interview 2, leading to loss of surrogates' data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 122 | 127
units on a scale | 0.8 [0.5 to 1.1] | 0.5 [0.2 to 0.8]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; Test type: Superiority; p < 0.05, generalized linear models — P values were calculated

6. Secondary Outcome: Quality of Communication Scale Score
Description: Here we report QOC score differences between Interview 1 (baseline) and Interview 2 (immediately post-intervention) for primary (not secondary) surrogate decision makers.
  Scores range from 0-110, with higher scores=better quality of communication.
Time Frame: Study day 1 (pre-randomization), ~2-7
Population: Note that the discrepancy between the number of surrogates in these analyses (122 and 127) differs from those enrolled (137 and 138). This is because the QOC requires complete data at both Interview 1 and Interview 2. Some patients died or regained decisional capacity before Interview 2, leading to loss of surrogates' data.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 122 | 127
units on a scale | 4 [1.3 to 6.8] | 7.0 [4.1 to 9.8]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; Test type: Superiority; p < 0.05, generalized linear models — P values were calculated

7. Secondary Outcome: Change in Clinical-surrogate Concordance Scale Score (Nurse)
Description: Concordance is calculated as the absolute value of the difference in prognosis for 1 year patient survival between the primary surrogate decision maker and the IUC nurse, and, therefore, can range from 0 to 100.
  We report pre-intervention to post-intervention difference in the CSCS.
  The CSCS is calculated as the absolute value of the difference between the surrogate's response and that of the nurse to the question, "What percent chance do you think [the patient/your loved one] has of being alive 1 year from now if the current treatment plan is continued?" Scores can range from 0 to 100 percentage points, and higher values indicate greater discordance.
Time Frame: ~2-7 days post-randomization
Population: nurses and primary surrogate decision makers
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Decision Aid | Usual Care
Number analyzed (Participants) | 94 | 101
units on a scale | -5.4 [-11.2 to 0.3] | -6.2 [-10.6 to -1.7]
Statistical Analysis 1: Comparison: Decision Aid vs Usual Care; To test the hypothesis, we used a general linear model fit with generalized estimating equations, a linear link, and an exchangeable correlation (PROC GENMOD). Model parameters included indictor variables for intervention, Interview 2, the interaction between intervention and Interview 2, and a 4-level site variable. The mean CSCS between-groups difference, corresponding 95% confidence interval (CI), and p value were derived from the intervention-by-Interview 2 interaction term; Test type: Superiority; p < 0.05, GEE — P values were calculated

ADVERSE EVENTS:
Time Frame: 6 months
Description: Collected on surrogates.
Arm/Group | Decision Aid | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/206
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/206
Other Adverse Events (participants affected / at risk) | 0/210 | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No